CLINICAL TRIAL: NCT04301648
Title: Impact in Quality of Care of the "STructural heARt NURSE" as New Interventional Cardiology Nursing Role in Spain. STAR Nurse Project.
Brief Title: Impact in Quality of Care of the "STructural heARt NURSE" as New Interventional Cardiology Nursing Role in Spain.
Acronym: STAR-Nurse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIBSP-STA-2019-123
Record Dates: First submitted 2020-03-03; First posted 2020-03-10 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Valvular Heart Disease; Nurse's Role; Competence; Cardiac Disease
Keywords: Quality of Health Care/organization & administration; Advanced Practice Nursing/trends; Quality Improvement/organization & administration; Quality of Health Care/standards; Professional Role; Structural Heart Disease; Nurse's Role; Valvular Heart Disease; Nurse's Competences
MeSH Terms: conditions — Heart Valve Diseases; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design study, pre-post intervention type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common Practice (Active Comparator): Patients included in the phase before will receive common practice.
  Interventions: Other: Common Practice
- STAR Nurse (Experimental): Patients included in the phase after will receive care by a STAR Nurse.
  Interventions: Other: STAR Nurse

INTERVENTIONS:
Other: STAR Nurse — This intervention will consist in that the nurse who is in the hemodynamic nurse's office will do the STAR Nurse's tasks and competences.
  Although the intervention will be detailed through phase 1 (integrative review) and 2 (Delphy methodology).
  It is expected that the main STAR nurse's competencies and tasks in the nurse's office will be:
  1. To guarantee a comprehensive evaluation and appropriate triage to candidates for an interventional procedure of structural heart disease, coordinating the request for complementary tests and previous visits.
  2. Make education to the patient and family.
  3. Make communication bridge with cardiologists.
  4. Establish specific patient-centered care processes.
  5. Promote continuity of care after discharge, follow up after discharge, and reevaluate quality of life and fragility.
  Arms: STAR Nurse
Other: Common Practice — Common practice will consist in that the nurse who is in the hemodynamic nurse's office will do her usual task that is exclusively health education.
  Arms: Common Practice

SUMMARY:
The hypothesis is that patients with structural heart disease who are treated by STructural heARt nurses obtain better results in indicators of quality of care, compared with the usual practice (or not assisted) by this type of new interventional cardiology's nursing role.

DETAILED DESCRIPTION:
Valvular disease is the future epidemic structural heart disease of developed countries. To slow or alter the course of the disease, cardiac valve repair or replacement is necessary. Transcatheter treatment has become a safe alternative to surgery. The United States and Canada developed the TAVI (Transcather Aortic Valve Implantation) program and TAVI Nurse is strongly supported by scientific societies as a key leadership role in the aortic stenosis care process. This nursing role is not implemented in Spain.

The objective of this study is to develop a new nursing role in interventional cardiology, similar to TAVI Nurse but including all the structural heart diseases, through conceptual definition and competencies, and evaluate its impact on the quality of care after of its implementation.

The new nursing role of a hemodynamics and interventional cardiology unit in Spain will be based on the model existing in other countries.

This study consists of three phases:

Phase I) Integrative review to explore and identify the definition and competencies of TAVI Nurse or another similar figure outside Spain, as well as identify quality of care indicators.

Phase II) The competences of these nurses will be contextualized in Spain, and indicators of quality of care will be defined through the consensus of experts using a Delphi methodology.

Phase III) Quasi-experimental pre / post study to assess the quality of care, through the indicators developed, of the implementation of the new nursing role.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) who have been or will undergo any procedure of structural heart disease in the hemodynamic and interventional cardiology unit of the Hospital de la Santa Creu i Sant Pau.
* Patients who accept to participate in the study.

Exclusion Criteria:

* Patients with cognitive impairment, mental disability or other serious difficulty communicating.
* Patients with insufficient fluency of the main languages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Structural Quality Indicators | 30 days
  Structural quality indicators developed through phase 1 (Integrative Review) and phase 2 (Delphi Methodology) results. However, it is expected that the main STAR nurse's structural quality indicators could be some like:
  - Percutaneous/transcatheter treatment waiting time (days). Data will be collected by medical history review.
Process Quality Indicators | 30 days
  Process quality indicators developed through phase 1 (Integrative Review) and phase 2 (Delphi Methodology) results. However, it is expected that the main STAR nurse's process quality indicators could be some like:
  - Evaluation of procedural risk (points). The Society of Thoracic Surgery (STS) risk score will be used.
  The classification of the results is:
  * Less than or equal to 2 points means low surgical risk.
  * From 3 to 5 points means intermediate surgical risk.
  * Upper than or equal to 6 means high surgical risk.
Outcome Quality Indicators | 30 days
  Outcome quality indicators developed through phase 1 (Integrative Review) and phase 2 (Delphi Methodology) results. However, it is expected that the main STAR nurse's outcome quality indicators could be some like:
  - Mortality after Percutaneous/transcatheter treatment for any medical cause (days). Data will be collected by medical history review.

CONTACTS AND LOCATIONS:
Locations (1):
- FGS Hospital de la Santa Creu i Sant Pau, Barcelona, Spain